CLINICAL TRIAL: NCT02596373
Title: A Randomized, Open-label, Positive-controlled, Single-institutional, Phase Ⅱ of Mitoxantrone Hydrochloride Liposome Injection in Advanced Recurrent or Metastatic Breast Cancer
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in Advanced Recurrent or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-HE1506/PRO/Ⅰ
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Advanced Recurrent or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Mitoxantrone Hydrochloride Liposome Injection 20 mg/m2 will be infused intravenously once over 1 hours in 250 ml 5％ glucose injection on the first day during a treatment phase of 4 weeks
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Mitoxantrone Hydrochloride Injection (Active Comparator): Mitoxantrone Hydrochloride Injection 14 mg/m2 will be infused intravenously once over 30 minutes in 150 ml 5％ glucose injection on the first day during a treatment phase of 4 weeks
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection

SUMMARY:
The hypothesis of this clinical research study is to discover if the study drug Mitoxantrone Hydrochloride Liposome Injection can shrink or slow the growth of advanced recurrent or metastatic breast cancer

DETAILED DESCRIPTION:
Mitoxantrone Hydrochloride Liposome Injection is a kind of anthraquinone compounds, and its antineoplastic effect has been viewed in preclinical tests. The investigator's phase Ⅰstudy has shown that the drug's toxicity is manageable and the tolerable does is 20 mg/m2. The hypothesis of this clinical research study is to discover if the study drug Mitoxantrone Hydrochloride Liposome Injection can shrink or slow the growth of advanced recurrent or metastatic breast cancer. The safety of Mitoxantrone Hydrochloride Liposome Injection will also be studied. Patients physical state, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if Mitoxantrone Hydrochloride Liposome Injection is safe and effective in advanced recurrent or metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to study specific screening procedures;
* ≥ 18 and ≤ 75 years of age,female;
* Advanced recurrent or Metastatic breast cancer, comfirmed by histological analysis and/or cytology analysis. Have failed for at least two chemotherapy regimen aimed to the advanced recurrent or metastatic focus;
* Adapted to receive chemotherapy;
* Women diagnosed with human epidermal growth factor receptor negative(HER2-); Women diagnosed with HER2+, and unable to be treated by Anti-HER2+ targeted therapy. HER2- is defined as 0 or 1+ staining on immunohistochemistry or FISH negative for gene amplification. HER2+ is defined as +++ staining on immunohistochemistry or FISH positive for gene amplification;
* Not suitable for endocrine theapy or tolerance to endocrine therapy;
* Have at least one measurable site of disease according to RECIST1.1 criteria;
* If chemotherapy regimens containing anthracycline-based drugs, duration from palindromia to this chemotherapy regimens is not less than 12 mounths;
* ECOG performance status of 0-2, life expectancy of more than 3 mounths;
* Cardiac function is almost normal(NYHA classification is Grade 1, LVEF≥ 50％);
* Sexually active women of childbearing potential must use a medically acceptable form of contraception;
* Adequate hepatic, renal and hematologic functions: leukocyte≥3.0×10^9/L,neutrophils≥1.5×10^9/L,platelets≥75×10^9/L, hemoglobin≥90g/L, serum bilirubin≤1.5×ULN, ALT≤2.5×ULN(5×for liver metastasis),AST≤2.5×ULN(5×for liver metastasis), creatinine clearance rate≤1.5×ULN;

Exclusion Criteria:

* Suffering from serious internal disease, including serious heart attack, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer;
* Uncontrolled brain metastases;
* Pregnant or lactating women;
* Mitoxantrone has been used before;
* Anthracycline-based drugs was used after relapse and metastasis;
* The cumulative doses of doxorubicin and epirubicin before inclusion have surpassed 360 mg/m2 and 600 mg/m2, respectively;
* Less than 4 weeks from the last chemotherapy, less than 4 weeks from the last radiotherapy, less than 2 weeks from the last endocrinotherapy; Other antineoplastic drugs need to be used in this study;
* History of anthracycline-based drug allergy;
* History of liposome drug allergy;
* Uncontrolled psychosis or uncontrolled infections disease;
* Unsuited to participate in thsi study judged by investigators;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective reponse rate) | 4-8 Months

SECONDARY OUTCOMES:
PFS(Progression free survival) | 2.5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Ph.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Wang L, Cao J, Li C, Wang X, Zhao Y, Li T, Du Y, Tao Z, Peng W, Wang B, Zhang J, Zhang S, Wang Z, Hu X. Efficacy and safety of mitoxantrone hydrochloride liposome injection in Chinese patients with advanced breast cancer: a randomized, open-label, active-controlled, single-center, phase II clinical trial. Invest New Drugs. 2022 Apr;40(2):330-339. doi: 10.1007/s10637-021-01182-7. Epub 2021 Oct 11. PMID 34633576